CLINICAL TRIAL: NCT02993835
Title: Iron Bioavailability From Fortified Food in Healthy Women
Brief Title: Iron Bioavailability From Fortified Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16.15.NRC
Record Dates: First submitted 2016-12-07; First posted 2016-12-15 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Iron Bioavailability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Labeled iron salt (Fe54) (Active Comparator): Labeled iron salt (Fe54) with bouillon
  Interventions: Other: Labeled iron salt Fe54
- Labeled iron salt (Fe57) (Active Comparator): Labeled iron salt (Fe57) with bouillon
  Interventions: Other: Labeled iron salt Fe57
- Labeled iron salt (Fe58) (Experimental): Labeled iron salt (Fe58) with bouillon
  Interventions: Other: Labeled iron salt Fe58

INTERVENTIONS:
Other: Labeled iron salt Fe54 — Fe salt enriched with Fe 54 isotopes
  Arms: Labeled iron salt (Fe54)
Other: Labeled iron salt Fe57 — Fe salt enriched with Fe 57 isotopes
  Arms: Labeled iron salt (Fe57)
Other: Labeled iron salt Fe58 — Fe salt enriched with Fe 58 isotopes
  Arms: Labeled iron salt (Fe58)

SUMMARY:
Determination of fractional iron absorption from bouillon fortified with 3 labeled iron compounds.

DETAILED DESCRIPTION:
This single center trial will be single-blind to the subject, controlled, fully randomized with crossover design in 22 healthy females aged 18-40 years old.

Subjects will attend 8 visits. At screening (V0), 3 consecutive feeding days (V1-V3), 14 days after last stable isotope intake again 3 consecutive feeding days (V4-V6), and 14 days after last stable isotope intake blood sampling (V7).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-40 years old
2. Healthy, based on the medical screening visit including a blood formula
3. Normal BMI for age (18.5-25.0 kg/m2)
4. Weight less than 65 kg
5. Able to understand and to sign written informed consent prior to trial entry
6. Informed consent signed

Exclusion Criteria:

1. Anemia or polycythemia respectively evidenced by one of the following criteria from a standard blood formula: number of erythrocytes 4.0 - 5.8 1012/l or Hb 120-160 g/l or Ht 35-55%. Subjects outside of this range will be excluded.
2. Significant blood losses over the past 6 months (i.e. trauma, major surgery, blood donation and other causes to be appreciated by the investigator).
3. Serum ferritin above 80 µg/L range. As a result, hemochromatosis will be excluded.
4. Any therapy or medication taken for any infectious and inflammatory disease in the past two weeks.
5. Relevant digestive (intestinal, gastric, hepatic or pancreatic), renal, metabolic disease, as determined by the screening visit and by self-report from the subjects.
6. Diagnosed food allergy.
7. Pregnancy (tested in plasma at screening) and/or lactation.
8. History of cancer within the past year.
9. Significant weight loss during the last 3 months (10% and more)
10. Any medication or supplement which may impact erythrocytes, Hb or Ht (to the opinion of the investigator).
11. Iron supplementation therapy or perfusion in the last three months.
12. Smokers (> 5 cigarettes per day).
13. Have a high alcohol consumption (more than 2 drinks/day).
14. Consumption of illicit drugs (anamnesis only).
15. Subject having a hierarchical link with the investigator or co-investigators.
16. Subject who cannot be expected to comply with treatment or study procedure.
17. Currently participating or having participated in another clinical trial during the past month prior to the beginning of this study.
18. Subjects not willing and/or not able to comply with scheduled visits and the requirements of the study protocol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Relative iron bioavailability (RBV) of 58Fe salt to 54Fe salt (i.e. FIA of 58Fe salt divided by FIA of 54Fe salt), RBV of 57Fe salt to 54Fe salt and RBV of 58Fe salt to 57Fe salt. The determination of FIA is a prerequisite for this calculation. | 14 days after last stable isotope adminstration
  FIA will be calculated based on the measured shift of iron isotope ratios in the blood 14 days after the test meal administrations. The amounts of 57Fe, 54Fe and 58Fe in the blood will be calculated on the principle of isotope dilution by considering that iron isotopic labels are not mono-isotopic (Walczyk et al., 1997; Cercamondi, 2013). Circulating iron will be calculated based on blood volume and hemoglobin concentration (Kastenmayer et al., 1994). Blood volume will be indirectly measured based on height and weight and calculated using the formula proposed by Brown et al (1962). For calculations of fractional absorption, 80% incorporation of the absorbed iron into red blood cells is assumed.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — ETH Zurich, Human Nutrition Laboratory
Locations (1):
- ETH Zurich, Human Nutrition Laboratory, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No